CLINICAL TRIAL: NCT02416986
Title: Effects of Smoking Environment on Craving and Smoking: A Pilot Study
Brief Title: Effects of Smoking Environment on Craving and Smoking
Acronym: CC2pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00056221; R01DA038442-01 (NIH)
Record Dates: First submitted 2015-04-08; First posted 2015-04-15 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-08

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: 6 hour smoking abstinence
Behavioral: Delay to Smoking Task (smoking cues) — Participants will be presented with an unlit cigarette of their brand and an opportunity to initiate ad lib smoking at any time during the 60-minute task. During this period, participants will be allowed to read books or magazines, but will hear a tone alerting them to view cues (standard smoking environments) for the final minute of each 6-minute period. A monetary reinforcer will be provided for each 6-minute period that a participant resists smoking. Once participants stop the task they can choose to smoke as much or a little as they want for the next 30 minutes. Participants will be provided with a smoking tab. Each cigarette they light will cost them from their tab.
Behavioral: Delay to Smoking Task (nonsmoking cues) — Participants will be presented with an unlit cigarette of their brand and an opportunity to initiate ad lib smoking at any time during the 60-minute task. During this period, participants will be allowed to read books or magazines, but will hear a tone alerting them to view cues (standard nonsmoking environments) for the final minute of each 6-minute period. A monetary reinforcer will be provided for each 6-minute period that a participant resists smoking. Once participants stop the task they can choose to smoke as much or a little as they want for the next 30 minutes. Participants will be provided with a smoking tab. Each cigarette they light will cost them from their tab.

SUMMARY:
The goal of this study is to evaluate the effects of exposure to standard smoking environments on ability to resist smoking as measured with a Delay to Smoking Task. The results of this study will inform whether the Delay to Smoking Task is a sensitive measure for evaluating environment-provoked craving and smoking behavior.

DETAILED DESCRIPTION:
Adult smokers (n=25) will complete 4 visits and a 6 month follow-up phone call. Participants will complete a Delay to Smoking Task following 6 hours smoking abstinence. The task involves viewing pictures of smoking and non-smoking locations and participants will have the choice to smoke a cigarette at any time during the session. A monetary reinforcer will be provided for each 6-minute period that a participant resists smoking. Once participants stop the task they can choose to smoke as much or a little as they want for the next 30 minutes. Participants will be provided with a smoking tab. Each cigarette they light will cost them from their tab. Measurements of tobacco craving, emotion ratings, and nicotine withdrawal will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* generally healthy
* between the ages of 18 and 55
* smoking an average of 5 cigarettes per day for at least one year
* breath CO level > 8 ppm (if ≤ 8 ppm, then NicAlert Strip = 6)
* no interest in quitting smoking for the duration of time required for the experiment

Exclusion Criteria:

* inability to attend all required experimental sessions
* use of psychoactive medications
* use of smokeless tobacco
* current alcohol or drug abuse
* use of illegal drugs as measured by urine drug screen (excluding marijuana)
* current use of nicotine replacement therapy or other smoking cessation treatment
* Blood Alcohol Level (BAL) > 0.00
* use of other tobacco products or e-cigarettes more than 9 days in the past 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in self-report craving measured by the cue-exposure rating scale | at 0 minutes, +30 minutes, +60 minutes and following first cigarette
Difference in number of subjects who initiate smoking during the smoking cue Delay to Smoking Task compared to the nonsmoking cue Delay to Smoking Task | following start of Delay to Smoking Task, up to 60 minutes
  If participant initiates smoking a cigarette during the Delay to Smoking Task
Number of minutes to first puff | following start of Delay to Smoking Task, up to +60 minutes
  Number of minutes to first puff of cigarette will be recorded for participants that initiate smoking

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McClernon, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States